CLINICAL TRIAL: NCT02685410
Title: Formative Research for an HIV Videogame for Young Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1301011336
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: HIV Prevention; STI Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One Night Stan Pilot Testing Group (Experimental): The pilot testing of the One Nigh Stan prototype intervention will utilize 20 young black women aged 18-24 as participants.
  Interventions: Other: One Night Stan Prototype

INTERVENTIONS:
Other: One Night Stan Prototype — The One Night Stan prototype, will be a social network game with the goal of risk reduction and HIV/STI prevention in young black women.

SUMMARY:
As part of Yale's Play2Prevent (www.Play2Prevent.org) program to develop videogame-based interventions targeting risk reduction and prevention in youth and young adults, this study is designed to develop a paper prototype and intervention design manual of an online social-network game, One Night Stan, with the goal of risk reduction and HIV/STI prevention in young black women. The ultimate plan is to incorporate focus group participants input and feedback into the development of a conceptual model, intervention manual, and videogame intervention prototype. This prototype will then be tested using 20 participants and will utilize a pre-post design to evaluate the effectiveness of the program.

DETAILED DESCRIPTION:
The specific aims of this study are to:

Develop an online social network game for HIV/STI risk reduction and prevention by conducting a first set of focus groups with a total of 25 participants (5 focus groups with 5 participants each) in order to better understand preferences for online social network and gaming platforms, characteristics and design.

These collected data, established theoretical constructs, and the literature will be harnessed to develop a conceptual model for HIV/STI risk reduction and prevention in this specific population of women.

From the data collected and the new conceptual model, an intervention manual will be created that will incorporate a culturally and socially-tailored online social network game intervention paper prototype and design manual. In an iterative fashion, a second series of focus groups will be conducted (5 groups with 5 participants each for a total of 25 participants) to refine the intervention.

To pilot test the prototype intervention we will determine, in a pre-post design: (a) the intervention's acceptability and feasibility based on self-report data on the game experience and (b) preliminary evidence of the efficacy of the intervention collecting data on 1) HIV/STI knowledge 2) intentions/attitudes regarding condom use and HIV/STI partner testing 3) self-efficacy to insist on condom use and HIV/STI partner testing 4) self-efficacy and beliefs related to sexual risk behaviors, 4) perceived social norms, and 5) behaviors related to condom use and partner HIV/STI testing.

The focus of this registration record will be the participants and collected outcomes used to assess the prototype of the social network game. Assessments will be conducted at baseline, 2 weeks after playing the game and at 4 weeks post follow up.

ELIGIBILITY:
Inclusion Criteria:

* African-American race
* Female
* Ages 18 to 24 yeats

Exclusion Criteria:

* Failure to meet all inclusion criteria will exclude individuals from participation in the study

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-06-18 (Actual); Study Completion 2016-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Condom Use | 2 Weeks
  The program will be assessed by determining if an increase in the incidence of condom use by participants occurred after 2 weeks exposure to the program.
Overall Incidence of Risk Behaviors Associated with HIV/STI Transmission | 2 Weeks
  The program will be assessed by determining if a decrease in the incidence of risk behaviors associated with HIV/STI transmission by participants occurred after 2 weeks exposure to the program.

SECONDARY OUTCOMES:
Incidence of Condom Use | Baseline
  Measured as the incidence of condom use by participants at baseline.
Incidence of Condom Use | 4 Weeks
  Measured as the incidence of condom use by participants at baseline.
Overall Incidence of Risk Behaviors Associated with HIV/STI Transmission | Baseline
  Measured as the incidence of risk behaviors associated with HIV/STI transmission by participants.
Overall Incidence of Risk Behaviors Associated with HIV/STI Transmission | 4 Weeks
  Measured as the incidence of risk behaviors associated with HIV/STI transmission by participants.
Incidence of Vulnerability to Risky Sexual Behaviors | Baseline
  The program will be assessed by determining if a decrease in incidence of vulnerability to risk behaviors associated with HIV/STI transmission by participants occurred after 2 weeks exposure to the program.
Incidence of Vulnerability to Risky Sexual Behaviors | 2 Weeks
  The program will be assessed by determining if a decrease in incidence of vulnerability to risk behaviors associated with HIV/STI transmission by participants occurred after 2 weeks exposure to the program.
Incidence of Vulnerability to Risky Sexual Behaviors | 4 Weeks
  The program will be assessed by determining if a decrease in incidence of vulnerability to risk behaviors associated with HIV/STI transmission by participants occurred after 2 weeks exposure to the program.
HIV/STI Knowledge | Baseline
  Items from the validated instruments the HIV-KQ and STD-KQ were compiled into 12 item questionnaire measuring knowledge of HIV and STI's. These items are true/false responses in nature and the total score is based on the number of correct responses. The highest score possible is 12, which indicates superior knowledge of HIV/STI related information.
  The HIV Knowledge Questionnaire (18-item version) is a brief self-administered measure of the individual's HIV-related knowledge. (http://www.midss.org/content/hiv-knowledge-questionnaire-hiv-kq-18)SRB
  The STD-KQ is a comprehensive 27-item index that attempts to measure knowledge about sexually transmitted diseases. It is intended for use in research and applied settings (http://www.midss.org/content/sexually-transmitted-disease-knowledge-questionnaire-std-kq).
HIV/STI Knowledge | 2 Weeks
  Items from the validated instruments the HIV-KQ and STD-KQ were compiled into 12 item questionnaire measuring knowledge of HIV and STI's. These items are true/false responses in nature and the total score is based on the number of correct responses. The highest score possible is 12, which indicates superior knowledge of HIV/STI related information.
  The HIV Knowledge Questionnaire (18-item version) is a brief self-administered measure of the individual's HIV-related knowledge. (http://www.midss.org/content/hiv-knowledge-questionnaire-hiv-kq-18)SRB
  The STD-KQ is a comprehensive 27-item index that attempts to measure knowledge about sexually transmitted diseases. It is intended for use in research and applied settings (http://www.midss.org/content/sexually-transmitted-disease-knowledge-questionnaire-std-kq).
HIV/STI Knowledge | 4 Weeks
  Items from the validated instruments the HIV-KQ and STD-KQ were compiled into 12 item questionnaire measuring knowledge of HIV and STI's. These items are true/false responses in nature and the total score is based on the number of correct responses. The highest score possible is 12, which indicates superior knowledge of HIV/STI related information.
  The HIV Knowledge Questionnaire (18-item version) is a brief self-administered measure of the individual's HIV-related knowledge. (http://www.midss.org/content/hiv-knowledge-questionnaire-hiv-kq-18)SRB
  The STD-KQ is a comprehensive 27-item index that attempts to measure knowledge about sexually transmitted diseases. It is intended for use in research and applied settings (http://www.midss.org/content/sexually-transmitted-disease-knowledge-questionnaire-std-kq).
Subjective Sexual Norms | Baseline
  Subjective sexual intentions are measured using items from a questionnaire. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual norms. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the more positive one's sexual norms are perceived (with respect to HIV/STI transmission).
Subjective Sexual Norms | 2 Weeks
  Subjective sexual intentions are measured using items from a questionnaire. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual norms. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the more positive one's sexual norms are perceived (with respect to HIV/STI transmission).
Subjective Sexual Norms | 4 Weeks
  Subjective sexual intentions are measured using items from a questionnaire. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual norms. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the more positive one's sexual norms are perceived (with respect to HIV/STI transmission).
Sexual Intentions | Baseline
  Sexual intentions are measured using a 10 item scale. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual intentions. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the more positive one's intentions are perceived (with respect to HIV/STI transmission)..
Sexual Intentions | 2 Weeks
  Sexual intentions are measured using a 10 item scale. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual intentions. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the more positive one's intentions are perceived (with respect to HIV/STI transmission)..
Sexual Intentions | 4 Weeks
  Sexual intentions are measured using a 10 item scale. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual intentions. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the more positive one's intentions are perceived (with respect to HIV/STI transmission)..
Multi-dimensional Condom Attitudes Scale | Baseline
  The multi-dimensional condom attitudes scale (MCAS) was adapted for use in the study. The MCAS contains 25 items that assess attitudes toward condoms using 7-point Likert scales; higher scores indicate more favorable attitudes toward condoms. Sample items include: "Women think men who use condoms are jerks"; and "If a couple is about to have sex and the man suggests using a condom, it is less likely that they will have sex." Prior research confirmed that the scale is multidimensional, with a five-factor structure: (a) Reliability and Effectiveness, (b) Pleasure, (c) Identity stigma, (d) Embarrassment about Negotiation and Use, and (e) Embarrassment about Purchase (Helweg-Larsen & Collins, 1994). Each item uses a 5 point scale (5 = strongly agree) to assess condom attitudes. The average of the items is used, where a 5 would indicate a superior overall attitude concerning the construct being measured.
Multi-dimensional Condom Attitudes Scale | 2 Weeks
  The multi-dimensional condom attitudes scale (MCAS) was adapted for use in the study. The MCAS contains 25 items that assess attitudes toward condoms using 7-point Likert scales; higher scores indicate more favorable attitudes toward condoms. Sample items include: "Women think men who use condoms are jerks"; and "If a couple is about to have sex and the man suggests using a condom, it is less likely that they will have sex." Prior research confirmed that the scale is multidimensional, with a five-factor structure: (a) Reliability and Effectiveness, (b) Pleasure, (c) Identity stigma, (d) Embarrassment about Negotiation and Use, and (e) Embarrassment about Purchase (Helweg-Larsen & Collins, 1994). Each item uses a 5 point scale (5 = strongly agree) to assess condom attitudes. The average of the items is used, where a 5 would indicate a superior overall attitude concerning the construct being measured.
Multi-dimensional Condom Attitudes Scale | 4 Weeks
  The multi-dimensional condom attitudes scale (MCAS) was adapted for use in the study. The MCAS contains 25 items that assess attitudes toward condoms using 7-point Likert scales; higher scores indicate more favorable attitudes toward condoms. Sample items include: "Women think men who use condoms are jerks"; and "If a couple is about to have sex and the man suggests using a condom, it is less likely that they will have sex." Prior research confirmed that the scale is multidimensional, with a five-factor structure: (a) Reliability and Effectiveness, (b) Pleasure, (c) Identity stigma, (d) Embarrassment about Negotiation and Use, and (e) Embarrassment about Purchase (Helweg-Larsen & Collins, 1994). Each item uses a 5 point scale (5 = strongly agree) to assess condom attitudes. The average of the items is used, where a 5 would indicate a superior overall attitude concerning the construct being measured.
Sexual Risk Behavior Beliefs | Baseline
  The validated instrument the SRBBS was used to create items as part of a questionnaire. The Sexual Risk Behavior Beliefs and Self-Efficacy Scales (SRBBS; Basen-Engquist et al., 1996) taps into major constructs addressed within condom use theory (health belief model, theory of reasoned action, and social learning theory), and thus the current study results would easily extend to multiple theoretical approaches. The SRBBS contains 22 self-report, Likert-type items that assess five subscales of interest: condom use attitudes (e.g., I believe condoms should always be used if a person my age has sex), self-efficacy in using and obtaining condoms (e.g., How sure are you that you could use a condom correctly or explain to your partner how to use a condom correctly?), and barriers to condom use (e.g., I would feel uncomfortable carrying condoms with me).
Sexual Risk Behavior Beliefs | 2 Weeks
  The validated instrument the SRBBS was used to create items as part of a questionnaire. The Sexual Risk Behavior Beliefs and Self-Efficacy Scales (SRBBS; Basen-Engquist et al., 1996) taps into major constructs addressed within condom use theory (health belief model, theory of reasoned action, and social learning theory), and thus the current study results would easily extend to multiple theoretical approaches. The SRBBS contains 22 self-report, Likert-type items that assess five subscales of interest: condom use attitudes (e.g., I believe condoms should always be used if a person my age has sex), self-efficacy in using and obtaining condoms (e.g., How sure are you that you could use a condom correctly or explain to your partner how to use a condom correctly?), and barriers to condom use (e.g., I would feel uncomfortable carrying condoms with me).
Sexual Risk Behavior Beliefs | 4 Weeks
  The validated instrument the SRBBS was used to create items as part of a questionnaire. The Sexual Risk Behavior Beliefs and Self-Efficacy Scales (SRBBS; Basen-Engquist et al., 1996) taps into major constructs addressed within condom use theory (health belief model, theory of reasoned action, and social learning theory), and thus the current study results would easily extend to multiple theoretical approaches. The SRBBS contains 22 self-report, Likert-type items that assess five subscales of interest: condom use attitudes (e.g., I believe condoms should always be used if a person my age has sex), self-efficacy in using and obtaining condoms (e.g., How sure are you that you could use a condom correctly or explain to your partner how to use a condom correctly?), and barriers to condom use (e.g., I would feel uncomfortable carrying condoms with me).
Self-Efficacy in Sexual Risk Behaviors | Baseline
  The validated instrument the SRBBS was used to create an 11 item questionnaire. The Sexual Risk Behavior Beliefs and Self-Efficacy Scales (SRBBS; Basen-Engquist et al., 1996) taps into major constructs addressed within condom use theory (health belief model, theory of reasoned action, and social learning theory), and thus the current study results would easily extend to multiple theoretical approaches. The SRBBS contains 22 self-report, Likert-type items that assess five subscales of interest: condom use attitudes.
Self-Efficacy in Sexual Risk Behaviors | 2 Weeks
  The validated instrument the SRBBS was used to create an 11 item questionnaire. The Sexual Risk Behavior Beliefs and Self-Efficacy Scales (SRBBS; Basen-Engquist et al., 1996) taps into major constructs addressed within condom use theory (health belief model, theory of reasoned action, and social learning theory), and thus the current study results would easily extend to multiple theoretical approaches. The SRBBS contains 22 self-report, Likert-type items that assess five subscales of interest: condom use attitudes.
Self-Efficacy in Sexual Risk Behaviors | 4 Weeks
  The validated instrument the SRBBS was used to create an 11 item questionnaire. The Sexual Risk Behavior Beliefs and Self-Efficacy Scales (SRBBS; Basen-Engquist et al., 1996) taps into major constructs addressed within condom use theory (health belief model, theory of reasoned action, and social learning theory), and thus the current study results would easily extend to multiple theoretical approaches. The SRBBS contains 22 self-report, Likert-type items that assess five subscales of interest: condom use attitudes.
Condom Self-Efficacy | Baseline
  The Condom Use Self-Efficacy Scale (CUSES) assesses efficacy to purchase condoms, apply and remove them, and negotiate their use with partners; ample evidence exists for the reliability of the CUSES (Brafford & Beck, 1991). The 15-item CUSES (Brien et al., 1994; Brafford & Beck, 1991) measures condom use self-efficacy using 5-point Likert scales; higher scores indicate stronger percepts of condom use efficacy.
Condom Self-Efficacy | 2 Weeks
  The Condom Use Self-Efficacy Scale (CUSES) assesses efficacy to purchase condoms, apply and remove them, and negotiate their use with partners; ample evidence exists for the reliability of the CUSES (Brafford & Beck, 1991). The 15-item CUSES (Brien et al., 1994; Brafford & Beck, 1991) measures condom use self-efficacy using 5-point Likert scales; higher scores indicate stronger percepts of condom use efficacy.
Condom Self-Efficacy | 4 Weeks
  The Condom Use Self-Efficacy Scale (CUSES) assesses efficacy to purchase condoms, apply and remove them, and negotiate their use with partners; ample evidence exists for the reliability of the CUSES (Brafford & Beck, 1991). The 15-item CUSES (Brien et al., 1994; Brafford & Beck, 1991) measures condom use self-efficacy using 5-point Likert scales; higher scores indicate stronger percepts of condom use efficacy.
Sexual Communication | Baseline
  Sexual communication behaviors are measured using items from a questionnaire. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual communication. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the better one's sexual communication.
Sexual Communication | 2 Weeks
  Sexual communication behaviors are measured using items from a questionnaire. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual communication. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the better one's sexual communication.
Sexual Communication | 4 Weeks
  Sexual communication behaviors are measured using items from a questionnaire. Each item uses a 5 point scale (5 = strongly agree) to assess various facets of sexual communication. The average of the items is used, where an average of 5 would be the highest possible score. The higher a respondent's score is, the better one's sexual communication.

OTHER OUTCOMES:
Satisfaction with Game Play/Acceptability and Feasibility | 2 Weeks
  A questionnaire assessing satisfaction with the game will be included in the assessment of the program. It will use a Likert scale to capture agreement with questions measuring users' satisfaction with game play. A higher user's total score, the more favorable their overall attitude towards using the game.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly D Hieftje, PhD, Principal Investigator — Yale University; Lynn Fiellin, M.D., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No